CLINICAL TRIAL: NCT02384187
Title: The Effects of Oral Gabapentin Premedication on Postoperative Nausea and Vomiting and Early Postoperative Recovery Profile in Pediatric Patients Undergoing Adenotonsillectomy
Brief Title: Gabapentin Premedication and Adenotonsillectomy in Pediatric Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, heba mohamed nassar, lecturer of anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: N-47-2014
Record Dates: First submitted 2015-02-20; First posted 2015-03-10 (Estimated); Last update posted 2015-12-23 (Estimated); Status verified 2015-12

CONDITIONS: Post Operative Nausea and Vomiting (PONV); Adenotonsillectomy
Keywords: Gabapentin; PONV; Adenotonsillectomy; Pediatrics
MeSH Terms: conditions — Vomiting; Postoperative Nausea and Vomiting | interventions — Gabapentin; Premedication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group C (Placebo Comparator): Patients in this group will receive 0.3 ml/kg of a placebo solution identical in taste, shape and color to the study medication two hours before the induction of anesthesia.
  Interventions: Drug: placebo
- Group GAB (Experimental): Patients in this group will receive 0.3 ml/kg (16 mg/kg) oral gabapentin solution (Neurontin 50 mg/ml, Pfizer Pharmaceutical) as premedication two hours before the induction of anesthesia
  Interventions: Drug: Gabapentin as premedication

INTERVENTIONS:
Drug: Gabapentin as premedication — Patients will receive 0.3 ml/kg (16 mg/kg) oral gabapentin solution (Neurontin 50 mg/ml, Pfizer Pharmaceutical) as premedication two hours before the induction of anesthesia
  Arms: Group GAB
Drug: placebo — Patients will receive 0.3 ml/kg of a placebo solution identical in taste, shape and color to the study medication two hours before the induction of anesthesia.
  Arms: Group C

SUMMARY:
The frequent incidence of postoperative vomiting and severe pain in children undergoing adenotonsillectomy, may delay postoperative oral intake and increase the risk of dehydration. Postoperative nausea and vomiting (PONV) is of multi-factorial origin in this group of patients, with a reported incidence ranging from 23% to 73%.

There is growing evidence that the perioperative administration of gabapentinin in adults is beneficial for preoperative anxiolysis, postoperative analgesia, reduction of postoperative nausea and vomiting, and delirium.

Only few studies in literature explored the analgesic effects of preoperative gabapentin as premedication in pediatric population. However, the antiemetic effect of gabapentin in pediatric patients was not systematically investigated before.

ELIGIBILITY:
Inclusion Criteria:

* Aged (3-12)
* ASA physical status I or II
* Scheduled for adenotonsillectomy surgery in Abu Elrish Al-Mounira Hospital

Exclusion Criteria:

* Patients who have active infection
* Obstructive sleep apnea
* Cognitive impairment
* Abnormal bleeding profile
* Renal or hepatic dysfunction
* History of allergic reaction to study medications or chronic use of anti-consultants will be excluded.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV | over the first postoperative 6 hours
  The number of patient complaints of nausea and or vomiting will be recorded in the first 6 hours postoperatively

SECONDARY OUTCOMES:
Pediatric Anesthesia Behavior score (PAB) | within10 minutes before the child falls asleep.
  the score will be assessed during induction of anesthesia. The child will be scored 1 if Happy; 2 if Sad; and 3 if Mad.
Incidence and severity of postoperative delirium | up to 60 minutes after the end of the operation.
  Emergence agitation scores will be recorded every10 min for the first 60 minutes postoperatively
Duration of recovery | up to 60 minutes after the end of surgery.
  The extubation time will be the time interval from discontinuation of sevoflurane until removal of the endotracheal tube. The time to interaction will be the time from discontinuation of sevoflurane until verbal contact or response to commands.
Time to first request of postoperative rescue analgesics. | over the first postoperative 6 hours
  the time interval between the end of surgery and the first request to postoperative analgesia
Postoperative analgesic consumption | over the first postoperative 6 hours
Objective pain scale (OPS) | over the first postoperative 6 hours
  The objective pain scale will be assessed at 30 minutes, 2, 4 and 6 hours postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdulatif, Professor of Anesthesia, Study Chair — Cairo University
Locations (1):
- Kasr Al Ainy, Cairo, Egypt